CLINICAL TRIAL: NCT04235569
Title: Evaluation of Warfarin Initiation at 3mg Versus 5mg for Anticoagulation of Mechanical Mitral Valve Replacement Patients
Brief Title: Warfarin Initiation in Mechanical Mitral Valve Replacement Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarah Sabry Hashem (Other)
Responsible Party: Sponsor-Investigator, Sarah Sabry Hashem, Msc, Clinical Pharmacy, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11222
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Mitral Valve Disease
Keywords: warfarin; anticoagulation; mitral valve replacement
MeSH Terms: interventions — Warfarin; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): a group of 25 patients received 5mg Marevan ® tablets as initiation warfarin dose in combination of enoxaparin (Clexane® ) as a bridging agent.INR was monitored daily and dose adjustments were done to reach therapeutic INR range (2-3) at which the Enoxaparen was discontinued.Follow up was continued till first INR reading in therapeutic range.
  Bleeding events due to overanticoagulation were monitored through the follow up period.
  Interventions: Drug: Warfarin Sodium 5 MG; Drug: Enoxaparin Sodium 100 MG/ML Prefilled Syringe
- Group II (Experimental): a group of 25 patients received 3mg Marevan ® tablets as initiation warfarin dose in combination of enoxaparin (Clexane® ) as a bridging agent.INR was monitored daily and dose adjustments were done to reach therapeutic INR range (2-3) at which the Enoxaparen was discontinued.Follow up was continued till first INR reading in therapeutic range.
  Bleeding events due to overanticoagulation were monitored through the follow up period.
  Interventions: Drug: Warfarin Sodium 3 MG; Drug: Enoxaparin Sodium 100 MG/ML Prefilled Syringe

INTERVENTIONS:
Drug: Warfarin Sodium 5 MG — warfarin sodium 5mg tablets
  Other Names: Marevan 5mg
  Arms: Group I
Drug: Warfarin Sodium 3 MG — warfarin sodium 3mg tablets
  Other Names: Marevan 3mg
  Arms: Group II
Drug: Enoxaparin Sodium 100 MG/ML Prefilled Syringe — Clexane® Syringes 2,000 IU (20 mg)/0.2 ml solution for injection in pre-filled syringes.
  Clexane® Syringes 4,000 IU (40 mg)/0.4 ml solution for injection in pre-filled syringes.
  Clexane® Syringes 6,000 IU (60 mg)/0.6 ml solution for injection in pre-filled syringes.
  Clexane® Syringes 8,000 IU (80 mg)/0.8 ml solution for injection in pre-filled syringes.
  Dose was determined individually for each patient as 1mg/kg every 12 hours.
  Other Names: Clexane

SUMMARY:
A prospective, comparative study evaluating warfarin initiation in a dose of 3mg versus 5mg in mechanical mitral valve prostheses patients who received anticoagulation with warfarin with the use of enoxaparen as a bridging agent .Fifty patients were included and compared in terms of the primary outcome time to reach therapeutic INR range.Other outcomes includes proportion of patients who achieved the target INR of 2.0-3.0 between day 3 and day 5, total dose of enoxaparin required for bridging, safety related to both doses of anticoagulants used

DETAILED DESCRIPTION:
Inpatients of The Cardiovascular hospital who had undergone mitral heart valve replacement with a mechanical prosthesis and commencing warfarin were eligible for inclusion. Patients were included after they had newly undergone elective surgery for implantation of mechanical mitral heart valves, had commenced on warfarin, received enoxaparin as a bridging agent and had INR monitored for a minimum of 4 consecutive days after warfarin initiation.

A total of 50 consecutive MVR patients were recruited. Each was assigned to either the group I (25 patients) or the group II (25 patients) group. All patients received the conventional postoperative treatment including: Diuretics, beta-blockers, digoxin or heart rate-regulating calcium channel blockers and anticoagulation bridging therapy using LMWH according to the European Society of Cardiology (ESC) Guidelines for the management of MVR and antibiotic for 48hour after surgery according to the investigator's hospital's antibiotic protocol.

Baseline evaluation included demographics and history taking. After obtaining the informed consent, information including age, weight, height, smoking state, and other diseases e.g. hypertension, diabetes, hyperlipidemias, etc. were documented for each patient. Medication history in details, as well as the background cardiovascular treatment was considered.

Blood samples were withdrawn from patients for evaluation of INR. Complete blood count, kidney and liver function tests were performed as part of the routine admission care.

All patients were followed up daily post operative till reaching an in range INR value. All patients were observed daily for INR values and dose adjusted accordingly and also estimation of incidence and severity of bleeding complications was done.

ELIGIBILITY:
Inclusion Criteria:

* New mechanical mitral valve prostheses patients who will receive anticoagulation with warfarin with the use of enoxaparen as a bridging agent.

Exclusion Criteria:

* Pregnant or lactating women
* Renal disorder (GFR = 45< mL/min) or patients on renal dialysis
* Hepatic disorder (Child Pugh class B or C)
* Clinically significant active bleeding.
* Recurrent DVT or PE.
* Baseline INR >1.2
* Asian ancestry
* Cancer
* Impaired nutritional status
* Alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of warfarin initiating dose and the corresponding dosing schedule: Time to reach therapeutic INR range (TTR) | 4-16 days
  Time to reach therapeutic INR range (TTR):The time in days required for the patient from the start of warfarin initiation till reaching the therapeutic

SECONDARY OUTCOMES:
Evaluation of overanticoagulation | from 3 to 5 days
  Proportion of patients who achieved the target INR of 2.0-3.0 between day 3 and day 5
Anticoagulation Safety evaluation | from 4 to 16 days
  Incidence of major and minor bleeding events
Low Molecular Weight Heparin consumption | from 4 to 16 days
  The total dose of enoxaparin in mg that the patient received till discontinuation of bridging
The Overall cost evaluation | from 4 to 16 days
  total cost spent in LE during the follow up period calculated by the summation of the cost of treatment , cost of bleeding event management and cost of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M Saleh, MD, Study Director — Ain Shams University; Lamiaa M ElWakeel, PhD, Study Director — Faculty of pharmacy Ain Shams University; Marwa A Ahmed, PhD, Study Director — Faculty of pharmacy Ain Shams University; Sarah S Hashem, Msc, Principal Investigator — The Cardiovascular Hospital Ain Shams University
Locations (1):
- The Cardiovascular Hospital, Heliopolis, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suwanawiboon B, Kongtim P, Chinthammitr Y, Ruchutrakool T, Wanachiwanawin W. The efficacy of 3-mg warfarin initiating dose in adult Thai patients, who required long-term anticoagulant therapy. J Med Assoc Thai. 2011 Feb;94 Suppl 1:S225-31. PMID 21721451
- [Background] Roberts G, Razooqi R, Quinn S. Comparing Usual Care With a Warfarin Initiation Protocol After Mechanical Heart Valve Replacement. Ann Pharmacother. 2017 Mar;51(3):219-225. doi: 10.1177/1060028016676830. Epub 2016 Oct 26. PMID 27798318
- [Background] Dong L, Shi YK, Xu JP, Zhang EY, Liu JC, Li YX, Ni YM, Yang Q, Han T, Fu B, Chen J, Ren L, Wei SL, Chen H, Liu KX, Yu FX, Liu JS, Xiao MD, Wu SM, Zhang KL, Huang HL, Jiang SL, Qiao CH, Wang CS, Xu ZY, Zhou XM, Wang DJ, Ni LX, Xiao YB, Jiang SL, Zhang GM, Liang GY, Yang SY, Bo P, Zhong QJ, Zhang JB, Zhang X, Zhu YB, Teng X, Zhu P, Huang F, Xiao YM, Cao GQ, Tian H, Xia LM, Lu FL, Liu YQ, Liu DX, Xu H, Yuan Y, Li M, Chang C, Wu XC, Xu Z, Guo P, Bai YJ, Xue WB, Jiang XY, Na ZH, Zeng QY, Cai H, Wang YL, Xiong R, Jin S, Zheng XM, Wu D. [The multicenter study on the registration and follow-up of low anticoagulation therapy for the heart valve operation in China]. Zhonghua Yi Xue Za Zhi. 2016 May 24;96(19):1489-94. doi: 10.3760/cma.j.issn.0376-2491.2016.19.006. Chinese. PMID 27266493
- [Background] Bayliss A, Faber P, Dunning J, Ronald A. What is the optimal level of anticoagulation in adult patients receiving warfarin following implantation of a mechanical prosthetic mitral valve? Interact Cardiovasc Thorac Surg. 2007 Jun;6(3):390-6. doi: 10.1510/icvts.2007.152819. Epub 2007 Feb 9. PMID 17669876
- [Background] Yoon IK, Lee KE, Lee JK, Chang BC, Gwak HS. Adequate intensity of warfarin therapy for Korean patients with mechanical cardiac valves. J Heart Valve Dis. 2013 Jan;22(1):102-9. PMID 23610997
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Jul 11;70(2):252-289. doi: 10.1016/j.jacc.2017.03.011. Epub 2017 Mar 15. No abstract available. PMID 28315732
- [Background] Mahtani KR, Heneghan CJ, Nunan D, Bankhead C, Keeling D, Ward AM, Harrison SE, Roberts NW, Hobbs FD, Perera R. Optimal loading dose of warfarin for the initiation of oral anticoagulation. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD008685. doi: 10.1002/14651858.CD008685.pub2. PMID 23235665
- [Derived] Sabry S, El Wakeel LM, Saleh A, Ahmed MA. Comparison of Warfarin Initiation at 3 mg Versus 5 mg for Anticoagulation of Patients with Mechanical Mitral Valve Replacement Surgery: A Prospective Randomized Trial. Clin Drug Investig. 2022 Apr;42(4):309-318. doi: 10.1007/s40261-022-01137-7. Epub 2022 Mar 10. PMID 35274222